CLINICAL TRIAL: NCT00455416
Title: Dietary Intervention in Stage III/IV Follicular Lymphoma. Impact on Markers of Cell Proliferation, Apoptosis, Host Immune Cell Infiltrate and Oxidative Stress.
Brief Title: Dietary Intervention in Follicular Lymphoma
Acronym: KLYMF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Harald Holte MD, PhD, Rikshospitalet-Radiumhospitalet HF
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dietary intervention FL
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2007-04

CONDITIONS: Follicular Lymphoma
Keywords: Low grade lymphoma; Diet; Antioxidants; Non Hodgkin Lymphoma - Follicular Lymphoma grade 1&2 stage III/IV
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acids; Selenium; allicin; Ellagic Acid; Resveratrol; Quercetin; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Omega 3 fatty acids (EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid)) — 1000mgx5 daily
  Other Names: Nycoplus omega-3 1000mg
Drug: Selenium (L-Selenomethionine), — 100mcgx2 daily
  Other Names: Solaray selenium 100mcg
Drug: Garlic extract (Allicin) — 6 garlic pearls daily
  Other Names: Circuline
Drug: Pomegranate juice (ellagic acid) — Pomegranate juice 100%, 660ml /495 ml every second day.
  Other Names: Produced by:Tine Meierier.
Drug: Grape juice (resveratrol, quercetin) — Merlot grape juice 100%, 660ml /495 ml every second day
  Other Names: Produced by Tine Meierier
Drug: Green Tea (Epigallocathechin gallate) — Green Tea. 2 cups daily
  Other Names: Green tea - twinings java green tea

SUMMARY:
A dietary intervention study in patients with Follicular Lymphoma (FL) Stage III/IV to assess the ability of several dietary factors to induce apoptosis, inhibit cell proliferation and modulate tumor cell infiltrate in vivo.

DETAILED DESCRIPTION:
Dietary factors plays an important role in the prevention of several diseases. The cardiovascular disease mortality have dropped dramatically the last 20 years, but the relative death rates from cancer remains fairly stable. There is reason to believe that factors in the tumors microenvironment is of great importance for the outcome of many malignant diseases, including FL. Factors predicting a poor outcome are associated with inflammation, oxidative stress which both impair the hosts immune response and produces growth stimulatory signals. In this open study with 45 patients to be included we seek to perform a dietary intervention with comparison of apoptosis rate, proliferation rate and immune cell infiltrate before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more.
* Permanent address in Norway, located in health region south or east. People living outside these areas in other health regions in Norway may be able to participate but after individual evaluation.
* Histologically verified follicular lymphoma grade I or II without clinical signs of transformation to aggressive lymphoma.
* Stage III/IV.
* Previously untreated or at least 1 year since rituximab treatment or 6 months since cytotoxic chemotherapy.
* Not scheduled for disease specific treatment for the next 3 months.
* At least one pathological superficial lymph node available for ultrasound guided biopsy.
* Cytologically and/or immunocytologically compatible with follicular lymphoma.
* Women with childbearing potential, only with use of safe contraceptives

Exclusion Criteria:

* Gross abnormalities in blood samples. (Hematologic values Hgb< 10, leukocytes< 2,5, trombocytes <100, liver enzymes (ALAT,ASAT,GT,ALP) > 2,5 x upper normal values,bilirubin >35 creatinine >130)
* Other serious medical illness (unstable cardiovascular disease, unstable pulmonary disease, uncontrolled diabetes, autoimmunity, chronic infection or other active cancer).
* Use of NSAID, ASA the last two weeks prior to enrollment.
* Use of systemic corticosteroids the last two months prior to enrollment.
* Regular use of anticoagulants as LMW Heparin or warfarin.
* Use of carbamazepin, nifedipin and other drugs metabolized with CYP 3A4 where interaction might cause hazardous side effects which cannot be controlled with serum measurements or organ function monitoring.
* Inclusion in another clinical trial which involves medication or nutritional supplements.
* Use of complementary medicine/alternative medicine which includes high dose* vitamins or antioxidants/nutritional supplements 2 weeks prior to sampling procedures .
* Regularly use of omega 3 fatty acids more than 1g / day
* History of serious or unstable medical or psychiatric disorder.
* History of heavy alcohol consumption > 3 units / day.
* Pregnancy
* Individuals judged by the clinical investigator to be unable to follow instructions and procedures of the study.

(*high dose is defined as vitamins or antioxidant supplements exceeding what is present in regular multi-vitamin supplements covering regular RDAs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Apoptosis an proliferation rate in tumor cells, | At the end of intervention (week 16)

SECONDARY OUTCOMES:
Levels of: proinflammatory cytokines,tumor immune cell infiltrate | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Harald Jr. Holte, MD, PhD, Principal Investigator — RRHF Rikshospitalet Radiumhospitalet HF
Locations (1):
- RRHF RIkshospitalet Radiumhospitalet HF, Montebello, Oslo County, Norway